CLINICAL TRIAL: NCT03962855
Title: The Thromboxane Receptor Antagonist to Block the Effects of Non-Platelet Thromboxane Generation and Improve Endothelial Function (TRAP) Trial
Brief Title: Thromboxane Receptor Antagonist to Improve Endothelial Function
Acronym: TRAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeffrey Rade (Other)
Collaborators: American Heart Association (Other); Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Rade, Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMMS-TPRA-01
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases; Vascular Dilation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single center, prospectively randomized, double-blinded, placebo-controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ifetroban (Active Comparator): Ifetroban 250 mg oral capsule administered once daily for a minimum of 4 weeks.
  Interventions: Drug: Ifetroban Sodium
- Placebo (Placebo Comparator): Matching placebo administered once daily for a minimum of 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ifetroban Sodium — Ifetroban sodium 250 mg capsule once daily for 4 weeks
  Arms: Ifetroban
Drug: Placebo — Placebo arm to match Ifetroban Sodium once daily for 4 weeks.
  Arms: Placebo

SUMMARY:
This study evaluates whether addition of the thromboxane receptor antagonist to chronic aspirin therapy improves endothelial function and reduces non-platelet thromboxane generation in patients with established cardiovascular disease. Half of participants will receive ifetroban and the other half will receive matching placebo for the 4 week study period.

DETAILED DESCRIPTION:
Thromboxane is a prostaglandin produced in healthy individuals mainly in platelets, where it mediates platelet activation and vasoconstriction via binding to cellular thromboxane-prostanoid (TP) receptors. The cardioprotective effect of aspirin is due to suppression of platelet thromboxane generation and reactivity. Unfortunately 25-50% of patients with cardiovascular disease taking ASA continue to generate thromboxane from non-platelet sources, which significantly increases their risk of atherothrombosis and death. Evidence suggests that oxidative stress is a potent stimulus for thromboxane generation in endothelial cells that involves autocrine/paracrine signaling through the TP receptor. This clinical trial addresses the central hypothesis that vascular endothelial cells under oxidative stress are a major source of non-platelet thromboxane generation in patients with cardiovascular disease and that antagonism of the TP receptor will suppress its formation and improve endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-80 years of age with established cardiovascular disease
* Take >=81 mg daily of aspirin as part of their daily medical regimen
* Urine thromboxane B2 metabolites >1145 pg/mg creatinine on screening.
* Able to provide written consent and comply with protocol-specific procedures.

Exclusion Criteria:

* Chronic oral anticoagulation with a non-vitamin K antagonist.
* Anticipated change or interruption in aspirin therapy during the study period.
* ST segment myocardial infarction within the past 30 days.
* Cardiac surgery within the past 30 days.
* Stage 4-5 renal failure or on renal replacement therapy.
* An ongoing uncontrolled severe inflammatory condition.
* Pregnant,intending to become pregnant or breast feeding.
* Known ifetroban or aspirin sensitivity Inability to perform vascular testing.
* Participation in another investigational drug trial within 30 days of randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Rade, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ifetroban | Placebo
Started | 29 | 28
Completed | 29 | 23
Not Completed | 0 | 5
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ifetroban | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (10.2) | 62.4 (9.9) | 63 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 19 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 26 | 26 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Reactive Hyperemia Index (RHI)
Description: The change in Reactive Hyperemia Peripheral Index (RHI) as measured by Arterial Tonometry.
  The Reactive Hyperemia Index (RHI) is calculated as the ratio of post- to pre-occlusion peripheral arterial tone signals on the occluded side, normalized to the control side, and further adjusted for baseline vascular tone. RHI is automatically measured by the EndoPAT 2000 software. According to the manufacturer, an RHI value greater than 1.67 is considered normal, while a lower value indicates endothelial dysfunction and is associated with an increased risk of cardiovascular events.
Time Frame: Baseline to 4 weeks
Population: 5 participants were withdrawn from the placebo group
Measure: Median (Inter-Quartile Range); unit: percentage index change
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 29 | 23
percentage index change | -0.01 [-0.36 to 0.34] | 0.21 [-0.17 to 0.51]

2. Secondary Outcome: Change in Percent Flow-mediated Vasodilation (FMD)
Description: The measure is the change in flow-mediated vasodilation (FMD) as measured by Brachial vasoractivity
Time Frame: Baseline to 4 weeks
Population: 5 participants from the placebo group were withdrawn from the study
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 29 | 23
percentage | 11.36 [-7.93 to 61.36] | -15.83 [-28.71 to -2.52]

3. Secondary Outcome: Change in Urinary TXB2-M
Description: Urinary urinary TXB2-M measured by 11-dhTXB2 ELISA
Time Frame: Baseline to 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mg creatinine
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 29 | 23
pg/mg creatinine | 370.7 [11.6 to 884.8] | -210.9 [-895.1 to 85.7]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Ifetroban | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 3/28
Other Adverse Events (participants affected / at risk) | 18/29 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ifetroban (N=29) | Placebo (N=28)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecistitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Celulitis on the left foot and ankle (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound complication (edema, erythema, pain) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cardiac chest pain (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infaction (Cardiac disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ifetroban (N=29) | Placebo (N=28)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Fatigue (General disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
AST increased (Investigations) | 2 (2) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Epistaxis (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Nasal congestion (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pharyngitis (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (2) | 0 (0)
ALT increased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Situational syncope (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alcohol Intolerance Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anemia (General disorders) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Leucocytosis (Immune system disorders) | 0 (0) | 1 (1)
Lymphocytopenia (Immune system disorders) | 0 (0) | 1 (1)
Neutrophilia (Infections and infestations) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical and medical procedure (Surgical and medical procedures) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT03962855/Prot_SAP_000.pdf